CLINICAL TRIAL: NCT01918605
Title: Protection of Rectum From High Radiation Doses During Prostate Cancer Low-dose Brachytherapy Using Diluted or Non-diluted DuraSeal as a Spacer
Brief Title: Protection of Rectum From High Radiation Doses Using a Spacer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Markku Vaarala, MD, PhD, Associate Chief Urologist, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OY-111
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site
Keywords: prostate cancer; brachytherapy; spacer; side effect
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diluted spacer (Experimental): Single dose of DuraSeal product with DuraSeal components diluted 1:1 in sterile saline injected between rectum and prostate
  Interventions: Device: Diluted spacer
- Non-diluted spacer (Active Comparator): Single dose of DuraSeal product injected between rectum and prostate
  Interventions: Device: Non-diluted spacer

INTERVENTIONS:
Device: Diluted spacer
  Other Names: DuraSeal
  Arms: Diluted spacer
Device: Non-diluted spacer
  Other Names: DuraSeal
  Arms: Non-diluted spacer

SUMMARY:
The purpose of this study is to evaluate the usefulness of diluted and non-diluted DuraSeal product as a spacer between prostate and rectum in prostate cancer low-dose brachytherapy.

DETAILED DESCRIPTION:
Radiation therapy for prostate cancer leads to inappropriate radiation dose to the rectum wall leading rectum adverse effects in long term for some patients. A resorbable spaces between prostate and rectum could decrease the incidence of these side effect. In this trial, men with prostate cancer with intention to curative treatment by low-dose brachytherapy will be recruited. The subjects will be randomized to receive either diluted or non-diluted DuraSeal product as a spacer between prostate and rectum. Diluted or non-diluted DuraSeal will be applied between rectum and prostate at the end of the brachytherapy seed implantation procedure. After the implantation of the brachytherapy seeds, a needle is placed between rectum and prostate through perineal skin under transrectal ultrasound guidance. The proper position of the needle is confirmed by the injection of 10-15 ml sterile saline solution. After that, DuraSeal components are diluted in 1:1 with sterile saline and 6-10 ml of this diluted product will be injected using DuraSeal applicator. If the subject is randomized to receive non-diluted DuraSeal, the procedure will be identical with the exception the DuraSeal components will not be diluted. The resolution of the spacer will be followed by repeated plain computer tomography (CT) of pelvis performed a day before operation, a day after the operation, and 4, 8 and 12 weeks after the operation. In addition, magnetic resonance imaging of pelvis performed 12 weeks after the operation. The space created between prostate and rectum will be documented by plain CT and magnetic resonance imaging. Rectum radiation dose will be calculated based on these scans. Time to DuraSeal resolution will be evaluated from the scans. Possible side effects will be collected by subject interviews during follow-up visits at 4, 8 and 12 weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer patients with planned low-dose brachytherapy for the treatment of prostate cancer

Exclusion Criteria:

* not willing to participate this study

Ages: 50 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in spacer volume | 1 day, 4 weeks, 8 weeks, 12 weeks
  Time to spacer resolution will be measured based on the distance between rectum wall and prostate on CT scans before operation and on defined time frame. In addition, magnetic resonance imaging of pelvis will be performed 12 weeks after the operation in order to confirm the extent of spacer.

SECONDARY OUTCOMES:
Side effects | 1 day, 4 weeks, 8 weeks, 12 weeks
  Possible side effects will be collected by subject interview and physical examination on specified time frame.
Rectum radiation dose | 1 day, 4 weeks, 8 weeks, 12 weeks
  Rectum dose will be calculated based on CT scans after brachytherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Markku Vaarala, MD,PhD, Principal Investigator — Oulu University Hospital; Merja Korpela, MD, Study Chair — Oulu University Hospital; Vesa-Pekka Heikkilä, PhL, Study Chair — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland